CLINICAL TRIAL: NCT03956472
Title: Can Osteopathy and Expiratory Resistance be Used in Prevention and/or Treatment of Acute Mountain Sickness ? a Randomized Controlled Field Study
Brief Title: Alternative Treatments in Acute Mountain Sickness
Acronym: TAIA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of european funding
Sponsor: Institut de Formation et de Recherche en Médecine de Montagne (Other)
Responsible Party: Principal Investigator, Hugo Nespoulet, Head of research, Institut de Formation et de Recherche en Médecine de Montagne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TAIA
Record Dates: First submitted 2016-11-16; First posted 2019-05-20 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Acute Mountain Sickness
Keywords: Altitude; Acute mountain sickness; Osteopathy; End expiratory pressure
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Osteopathic group (Experimental): LCS Drainage before altitude exposure
  Interventions: Procedure: Osteopathic protocol for improving drainage of LCS; Other: PEEP-Sham
- PEEP 10 cmH2O (Experimental): 10 min at rest
  Interventions: Device: PEEP 10cmH2O; Other: Fake Osteopathic protocol
- Control group (Sham Comparator): Sham PEEP and fake osteopathic protocol
  Interventions: Other: Fake Osteopathic protocol; Other: PEEP-Sham

INTERVENTIONS:
Procedure: Osteopathic protocol for improving drainage of LCS — Osteopathic intervention improving drainage of LCS and cerebral blood flow through opitmizing veinous circulation
  Arms: Osteopathic group
Device: PEEP 10cmH2O — Breathing through a 10 cmH2O expiratory resistance for 10 min every 2 hours during 10h at 3842m high
  Arms: PEEP 10 cmH2O
Other: Fake Osteopathic protocol — Placebo intervention
  Arms: Control group; PEEP 10 cmH2O
Other: PEEP-Sham — PEEP 0 cmH2O (hidden)
  Arms: Control group; Osteopathic group

SUMMARY:
The purpose of this research is to support a hypothesis that osteopathic manual medicine (OMM) and / or a 10 cmH2O end-expiratory pressure (PEEP) could be used in the prevention of acute mountain sickness (AMS).

During altitude exposure, an exaggerated hypoxemia and the increase of intracranial pressure are both known to be major physipathological ways of AMS development.

The goal of the osteopathic protocol is to release tension on the circulatory structures directly related to cranial circulation and drainage. The main hypothesis is that it could lead to lower intracranial pressure and help reducing AMS signs. Furthermore the investigators would like to define a osteopathic score for individual AMS sensitivity, based on cranial bones mobility.

Several studies have shown that using PEEP at altitude (or hypoxia) increases SpO2. As for osteopathy protocol, the investigators would like to apply this experimental condition during real altitude exposure in a randomized controlled protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Experienced alpinist
* No previous acclimatization

Exclusion Criteria:

* Heart failure, respiratory failure, kidney failure
* Pregnant woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in Lake Louise Score from baseline to altitude continuous exposure. | mesured and reported every hour during a 10 hours altitude exposure
  Signs of acute mountain sickness regarding its severity according the official Lake Louise Score.

SECONDARY OUTCOMES:
Changes in numeric scale of well being from baseline to altitude continuous exposure. | every hour during a 10 hours altitude exposure
  Quantification of general feeling on a scale from 0 (feeling as before ascent) to 10 (worst feeling)

CONTACTS AND LOCATIONS:
Locations (1):
- Ifremmont, Chamonix, France